CLINICAL TRIAL: NCT03167931
Title: Neuromodulation by Non-invasive Brain Stimulation (NEUROMOD)
Brief Title: Neuromodulation by Non-invasive Brain Stimulation
Acronym: NEUROMOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 38RC17.078; 2017-A00834-49 (Other: ansm)
Record Dates: First submitted 2017-04-18; First posted 2017-05-30 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Healthy; Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation
Keywords: non-invasive brain stimulation; neuromodulation; semantic tasks
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: outcoume measure comparison is done between both age groups (18-49 years and 50-85 years).
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant is included for 2 neuromodulation sessions: one session where neurostimulation is effective, one session where neurostimulation is simulated. Sessions are performed blind for the participant and the outcome assessor.
  Sessions order is randomized for each participant (no arm randomization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18-49 years group (Experimental): Participants undergo 2 sessions of MRI + transcranial Magnetic Stimulation or transcranial electric stimulation + electroencephalogram. The 2 sessions are performed with an interval of 3 to 7 days.
  Interventions: Other: MRI + transcranial Magnetic Stimulation; Other: transcranial electric stimulation + electroencephalogram
- 50-85 years group (Experimental): Participants undergo 2 sessions of MRI + transcranial Magnetic Stimulation or transcranial electric stimulation + electroencephalogram. The 2 sessions are performed with an interval of 3 to 7 days.
  Interventions: Other: MRI + transcranial Magnetic Stimulation; Other: transcranial electric stimulation + electroencephalogram

INTERVENTIONS:
Other: MRI + transcranial Magnetic Stimulation — Healthy subjects undergo 2 sessions of MRI + transcranial Magnetic Stimulation + transcranial electric stimulation + electroencephalogram. The 2 sessions are performed with an interval of 3 to 7 days.
Other: transcranial electric stimulation + electroencephalogram — Healthy subjects undergo 2 sessions of MRI + transcranial Magnetic Stimulation + transcranial electric stimulation + electroencephalogram. The 2 sessions are performed with an interval of 3 to 7 days.

SUMMARY:
The main objective of this study is to estimate the effect of the neuromodulation on the behavioral performances during the access in semantics according to the age of the individuals.

Neuromodulation by non-invasive stimulation allows to explore the functioning of the brain by exciting or by inhibiting localized cortical zones. The modulation of the performances in cognitive tasks, further to the neuromodulation of these zones, allows to deduce on their functional roles.

DETAILED DESCRIPTION:
The objective of this project is to determine the changes of behavioral performances (time of answer, percentage of correct answers) further to the neuromodulation. The specific question is to estimate the effect on the performances of access at the semantic representations of this method, according to the age. One of the hypotheses in the research on the normal ageing is the difficulty of access to these representations (fundamental process for the cognitive functions, such as the language and the memory) at the healthy elderly. By using the neuromodulation the investigators wish to explore this hypothesis and to understand if the neuromodulation can have a beneficial effect on the improvement of the behavioral performances of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Major healthy Subject ( 18 - 85 years)
* Right-hander
* Signed Informed consent
* A medical examination must be made before the participation for the research
* Membership in or beneficiary of a national insurance scheme

Non inclusion Criteria:

* Subject under age 18 and of more than 85 years.
* Contraindications in the practice of MRI, TMS and tES
* Existence of a severe affection on the general plan: cardiac, respiratory, hematological, renal, hepatic, cancerous
* Regular taking of anxiolytic, sedative, antidepressant, neuroleptic
* Characterized psychiatric pathology
* Ingestion of alcohol before the examination
* Pregnancy, parturiency or breast-feeding
* Private person of freedom by court or administrative order, nobody being the object of a legal protective measure (under guardianship or guardianship)
* Participation to other protocols of current search with period of exclusion or in the previous week
* Subject which would perceive more than 4500 euros of compensation because of its participation in other searches involving the human person in 12 months preceding this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Effect of the neuromodulation on the behavioral performances during the access in semantics | 3 hours
  Evaluation of the changes of the behavioral performances before and after the neuromodulation by non-invasive cortical stimulation according to the age. More exactly, the investigators shall compare response times before and after neuromodulation between both age groups (18-49 years and 50-85 years), by testing the interaction between the effect of the neuromodulation and the age.

SECONDARY OUTCOMES:
Estimate the effect of the neuromodulation on the behavioral performances | 3 hours
  Compare the percentages of correct answers before and after neuromodulation by non-invasive cortical electric stimulation, according to the age (18-49 years vs 50-85 years).
Estimate the effect of transcranial Electrical Stimulation (tES) on the cognitive performances by neuropsychological scores, according to the age. | 3 hours
  Comparison of the neuropsychological scores before and after tES, according to the age (18-49 years vs 50-85 years).
Estimate the effect of tES on the cerebral functional activity, by comparing blood-oxygen-level dependent (BOLD ) signal or functional MRI before and after tES according to the age (18-49 years vs 50-85 years). | 3 hours
  The investigators extract estimates parameters (Estimated Beta weight Values) corresponding to each tES stimulation. Each session is be designed by using general linear model (Friston, 1998, statistical parametrical mapping in fMRI) defined as Ybefore tES = R1Beta1+R2Beta2 +R0Beta0 + e and Yafter tES = R1Beta1 +R2Beta2 +R0Beta0 + e, with Y = acquired BOLD signal, e = error, R1Beta1 corresponding to the task (meaning interest activation) regressor and R2Beta2 corresponding to the control (meaning no interest activation) regressor respectively convolved with the canonical hemodynamic response function (cHRf) and R0B0 corresponding to the constant regressor. Parameter estimates are calculated by extracting Beta1 and Beta2 values for each session respectively in order to compute statistical comparison (measure by subject) on the outcome measure (Beta1 before tES - Beta1 after tES).
Estimate the effect of the Transcranial Magnetic Stimulation (TMS) on the cognitive performances by neuropsychological scores, according to the age. | 3 hours
  Comparison of the neuropsychological scores before and after Transcranial Magnetic Stimulation (TMS), according to the age (18-49 years vs 50-85 years).
Estimate the effect of the TMS on the intellectual functional activity, according to the age. | 3 hours
  Comparison of the cerebral functional activity (electric neuronal signal, EEG) before and after TMS, according to the age (18-49 years vs 50-85 years).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Grenoble, France

REFERENCES:
- [Background] Monti A, Ferrucci R, Fumagalli M, Mameli F, Cogiamanian F, Ardolino G, Priori A. Transcranial direct current stimulation (tDCS) and language. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):832-42. doi: 10.1136/jnnp-2012-302825. Epub 2012 Nov 8. PMID 23138766
- [Background] Liuzzi G, Freundlieb N, Ridder V, Hoppe J, Heise K, Zimerman M, Dobel C, Enriquez-Geppert S, Gerloff C, Zwitserlood P, Hummel FC. The involvement of the left motor cortex in learning of a novel action word lexicon. Curr Biol. 2010 Oct 12;20(19):1745-51. doi: 10.1016/j.cub.2010.08.034. Epub 2010 Sep 30. PMID 20888226
- [Background] Holland R, Leff AP, Josephs O, Galea JM, Desikan M, Price CJ, Rothwell JC, Crinion J. Speech facilitation by left inferior frontal cortex stimulation. Curr Biol. 2011 Aug 23;21(16):1403-7. doi: 10.1016/j.cub.2011.07.021. Epub 2011 Aug 4. PMID 21820308
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Zimerman M, Hummel FC. Non-invasive brain stimulation: enhancing motor and cognitive functions in healthy old subjects. Front Aging Neurosci. 2010 Dec 1;2:149. doi: 10.3389/fnagi.2010.00149. eCollection 2010. PMID 21151809